CLINICAL TRIAL: NCT02062554
Title: Brasilia Heart Study of Outcome Markers in ST-elevation Myocardial Infarction
Brief Title: Brasilia Heart Study
Acronym: BHS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Collaborators: University of Brasilia (Other)
Responsible Party: Principal Investigator, Andrei Carvalho Sposito, Professor PhD MD, University of Campinas, Brazil
Other Study IDs: BHS-1
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: ST-Elevation Myocardial Infarction
Keywords: Myocardial infarction; Clinical outcome; Flow-mediated dilation; Inflammation
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Plasma Leucocyte DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
BHS is a cohort study of consecutive myocardial infarction (MI) patients admitted within the first 24 hours of symptoms and has been ongoing since May of 2006. The purpose of this study is to assess for possible markers for increased risk after MI.

DETAILED DESCRIPTION:
In-hospital assessment Patients admitted into the study are being submitted to in-hospital evaluation and blood samples collection upon admission (D1) and at the fifth day (D5) of MI. Patients are treated according to current US guidelines for STEMI and assistant physicians are responsible for all medical decisions without any influence of the investigators. Plasma and DNA samples are aliquoted for storage at -80 °C. DNA is extracted using QIAamp DNA Blood Mini Kit (Quiagen, GmBH Hilden).

Follow-up After hospital discharge, patients are referred for a guideline-driven medical therapy at the study outpatient clinic and were reevaluated during visits every three months. Lifestyle counseling for diet, smoking cessation, regular physical activity and weight loss was oriented for all patients. Follow-up prescriptions include simvastatin with the addition of ezetimibe when necessary (LDL-C goal of 70 mg/dL), captopril or losartan for hypertension or reduced ejection fraction (<40%); hypoglycemic treatment to achieve a HbA1c goal ≤7% or 8% for individuals aged of 60 years or older; aspirin 100 mg/day and clopidogrel 75 mg/day; and anti-ischemic therapy as required (propranolol and isosorbide dinitrate, alone or in combination).The physicians involved in the clinical follow-up were blind to all the analysis performed in the study.

Biochemical analysis Blood plasma samples are assessed for the following: blood glucose (Glucose GOD-PAP, Roche Diagnostics, Mannheim, Germany), total cholesterol (CHOD-PAP, Roche Diagnostics, Mannheim, Germany), triglycerides (TG) (GPO-PAP, Roche Diagnostics, Mannheim, Germany), high-density lipoprotein cholesterol (HDL-C) (HDL cholesterol without sample pre-treatment, Roche Diagnostics, Mannheim, Germany), C-reactive protein (CRP) (high-sensitivity CRP, Cardiophase, Dade Behring, Marburg, Germany), 8-isoprostane (EIA kit, Cayman Chemical Company, Ann Arbor, MI, USA), interleukin-2 (IL-2) (Fluorokine® MAP Human IL-2 Kit, R&D Systems, Minneapolis, MN, USA), tumor necrosis factor type α (TNF-α) (Fluorokine MAP Human TNF-α Kit, R&D Systems), and HbA1c (Variant II, Bio-Rad Laboratories, Hercules, CA, USA). Low-density lipoprotein cholesterol (LDL-C) is calculated by the Friedewald formula. Plasma insulin and C-peptide concentrations were determined by electrochemiluminescence (Roche Diagnostics, Mannheim, USA) and by imunoquimioluminescence (Immulite 2000, Diagnostic Products Corporation, Los Angeles, CA, USA), respectively. The Homeostasis Model Assessment version 2 (HOMA2) is used to estimate β-cell function (HOMA2%β) and insulin sensitivity (HOMA2%S). We use fasting plasma insulin levels to compute HOMA2%S, and plasma C-peptide to compute HOMA2%β. To evaluate nitric oxide (NO) production, the plasma levels of nitrite and nitrate (NOx) are measured by an NO chemiluminescence analyzer (model NOA, Sievers Instruments, Boulder, CO) after reduction with acidic vanadium (III) chloride.

Brachial Artery Reactivity Brachial artery reactivity is assessed systematically 30 days (D30) after STEMI to estimate the decline in endothelial function that persists after the acute phase stress. At the time of the measurement, all patients are on the abovementioned secondary prevention protocol for at least 3 weeks, including simvastatin at the starting dose of 20 mg/day. Brachial artery measurements are performed after over-night fasting and any vasoactive medications were withdrawn 24 hours before assessment. After 10 minutes of rest in a quiet room with the temperature controlled around 22°C, the brachial artery is located above the elbow, and a longitudinal image of 6 to 8 cm was taken as the resting scan. A blood pressure cuff is placed on the forearm and inflated to 50 mm Hg above the systolic blood pressure for 5 min. The cuff is deflated, and the flow-mediated dilation (FMD) scan is obtained for two minutes. Ten minutes later, baseline measurements were repeated before and after five mg of isosorbide dinitrate. The percentage change in diameter for FMD and nitrate-mediated dilation was calculated in relation to the respective baseline scans. Brachial artery reactivity is analyzed by the same experienced physician who is blinded to the patients' data. The intra-observer reproducibility has been 95%.

Echocardiography All echocardiographic measurements are performed according to American Society of Echocardiography and European Association of Echocardiography recommendations. All subjects undergo complete 2D ECHO using standard ultrasound equipment (iE 33 system, 2-5MHz sector transducer; Philips Medical Systems, Andover, MA), at D30. Images are acquired with simultaneous electrocardiographic (ECG) monitoring. Images are stored in DICOM (Digital Imaging and Communication in Medicine) for further measurements "offline". Quantifications are performed by averaging of three measurements. For ventricular remodeling evaluation the following measures are performed: LV end-diastolic diameter (LVEDD), LV end-systolic diameter (LVESD), LV septum diastolic thickness (SD) and posterior wall diastolic thickness (PD). Left ventricular mass (LVM) is calculated formula Devereux formula and indexed to body surface area (LVMI). LV wall relative thickness (ER) is calculated using the formula (2 x PPD) / LVEDD). Left ventricle end diastolic volume (LVEDV) and systolic volume (LVESV) and LE ejection fraction (LVEF) are calculated using Simpson's method.

Carotid ultrasound The intima-media thickness (IMT) and the presence of carotid plaques are assessed using high-resolution ultrasound (Philips, Model IE 33, 3-9 MHz linear transducer, Philips Medical Systems, Andover, Massachusetts, USA) according to the protocols of the American Society of Echocardiography. The measurements are performed bilaterally in the posterior wall of the common carotid bulb and the internal carotid artery through an automatic edge detection program (QLAB version 6.0 software). The carotid plaque is defined as the presence of focal thickening of at least 50% higher than the adjacent areas or as a focal region with IMT ≥ 1.5 mm.

Coronary angiography Coronary angiography is systematically performed in all enrolled patients according to standard techniques. Lumen narrowing >70% is considered as a significant stenosis. All coronary angiographies are classified by the Gensini score method. Efficacy of reperfusion is estimated by TIMI flow grade and myocardial blush grade (MBG) in the first angiogram after thrombolysis or percutaneous coronary intervention. All angiographic data are obtained by consensus of two experienced interventional cardiologists who are blinded to the investigation data.

Cardiac Magnetic Resonance Imaging (CMRI) CMRI are performed at D30 and all patients are studied in supine position in a 1.5T scanner (Signa CV/i, General Electric Healthcare, Milwaukee, Wisconsin) with an 8-element cardiac phased-array surface receiver coil. All CMRI are acquired during breath-holds with ECG gating. LV size and function imaged by cine steady-state free-precession (typical TR 3.4 ms; TE 1.2 ms; temporal resolution 40-50 ms; in-plane spatial resolution 1.5-1.8 mm and 1.8-2.1 mm, depending on the field of view) are performed in multiple parallel short-axis planes (8 mm thick without spacing) and three radial long-axis planes. Using a previously described sequence[9] (repetition time, 4.8 ms; echo time, 1.3ms; in-plane spatial resolution between 1.5 X 2.0 mm and 1.9 X 2.0 mm), late gadolinium enhancement images (LGE) at matching cine-image slice locations are acquired 10 to 15 minutes after intravenous gadolinium-DTPA administration (0.15 to 0.20 mmol/kg; Magnevist, Berlex Pharmaceuticals, Wayne, NJ).

Statistical methods Categorical variables are compared by use of the chi-square test. Analysis of covariance (ANCOVA) is used to assess the association between the potential markers. Adjustments for baseline levels, age and gender are performed in all comparisons. Assumptions of the ANCOVA models (linearity, normality of distribution and equal variance) are checked using histograms, normal probability plots and residual scatter plots. Estimates of the cumulative event rate are calculated by the Kaplan-Meier method and the comparison between curves is made by Log rank test. For Cox multivariable regression models, the proportional hazard assumption is tested by adding time-dependent interaction variables that are confirmed to be valid in each of the models. A two-sided p-value of 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* less than 24 hours after the onset of MI symptoms
* ST-segment elevation of a least 1 mm (frontal plane) or 2 mm (horizontal plane) in two contiguous leads
* myocardial necrosis, as evidenced by increase to at least one value above the 99th percentile above the reference limit of CK-MB (25 U/L) and troponin I (0·04 ng/mL) followed by a decline of both

Exclusion Criteria:

* Cognitive impairment
* Patients unable to attend follow-up
* Concomitant diseases with short-term survival expectancy, i.e. cancer, severe COPD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ST-elevation Myocardial Infarction patients admitted to Hospital de Base de Distrito Federal, Brasilia, Brazil
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2006-05; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 30 days

SECONDARY OUTCOMES:
Major cardiovascular events | 2 years
  Sudden cardiac death (unrelated to trauma, unexpected, and occurring in less than six hours after onset of symptoms), fatal MI (any death preceded by MI) or non-fatal MI.
All cause mortality | 2 years

OTHER OUTCOMES:
Endothelial Function | 30 days
  Assessment of endothelial function on brachial artery. The flow-mediated dilation was measured.
Left Ventricular Remodeling | 30 days
  Left Ventricular (LV) Remodeling as indicated by LV end-diastolic diameter (LVEDD), LV end-systolic diameter (LVESD), LV septum diastolic thickness (SD) and posterior wall diastolic thickness (PD).

CONTACTS AND LOCATIONS:
Overall Officials: Andrei C Sposito, PhD MD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- State University of Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Result] Quinaglia e Silva JC, Coelho-Filho OR, Andrade JM, Quinaglia T, Modolo RG, Almeida BO, van der Geest RJ, Jerosch-Herold M, Coelho OR, Sposito AC; Brasilia Heart Study Group. Peri-infarct zone characterized by cardiac magnetic resonance imaging is directly associated with the inflammatory activity during acute phase myocardial infarction. Inflammation. 2014 Jun;37(3):678-85. doi: 10.1007/s10753-013-9784-y. PMID 24282109
- [Result] Figueiredo VN, Godoi FC, Martins NS, Quinaglia e Silva JC, Nadruz W Jr, Coelho OR, Sposito AC; Brasilia Heart Study Group. Diabetes mellitus unawareness is a strong determinant of mortality in patients manifesting myocardial infarction. Curr Med Res Opin. 2013 Nov;29(11):1423-7. doi: 10.1185/03007995.2013.832186. Epub 2013 Sep 4. PMID 23927444
- [Result] Carvalho LS, Martins NV, Moura FA, Cintra RM, Almeida OL, Quinaglia e Silva JC, Sposito AC; Brasilia Heart Study Group. High-density lipoprotein levels are strongly associated with the recovery rate of insulin sensitivity during the acute phase of myocardial infarction: a study by euglycemic hyperinsulinemic clamp. J Clin Lipidol. 2013 Jan-Feb;7(1):24-8. doi: 10.1016/j.jacl.2012.10.003. Epub 2012 Oct 26. PMID 23351579
- [Result] Costa AP, de Paula RC, Carvalho GF, Araujo JP, Andrade JM, de Almeida OL, de Faria EC, Freitas WM, Coelho OR, Ramires JA, Quinaglia e Silva JC, Sposito AC; Brasilia Heart Study Group. High sodium intake adversely affects oxidative-inflammatory response, cardiac remodelling and mortality after myocardial infarction. Atherosclerosis. 2012 May;222(1):284-91. doi: 10.1016/j.atherosclerosis.2012.02.037. Epub 2012 Mar 3. PMID 22436606
- [Result] Carvalho LS, Cintra RM, Moura FA, Martins NV, Quinaglia E Silva JC, Coelho OR, Sposito AC; Brasilia Heart Study Group. High plasma HDL-C attenuates stress hyperglycemia during acute phase of myocardial infarction. Atherosclerosis. 2012 Jan;220(1):231-6. doi: 10.1016/j.atherosclerosis.2011.09.044. Epub 2011 Oct 4. PMID 22018645
- [Result] Sposito AC, Alvarenga BF, Alexandre AS, Araujo AL, Santos SN, Andrade JM, Ramires JA, Quinaglia E Silva JC, Coelho OR; Brasilia Heart Study Group. Most of the patients presenting myocardial infarction would not be eligible for intensive lipid-lowering based on clinical algorithms or plasma C-reactive protein. Atherosclerosis. 2011 Jan;214(1):148-50. doi: 10.1016/j.atherosclerosis.2010.10.034. Epub 2010 Nov 3. PMID 21115179
- [Result] Sposito AC, Carvalho LS, Cintra RM, Araujo AL, Ono AH, Andrade JM, Coelho OR, Quinaglia e Silva JC; Brasilia Heart Study Group. Rebound inflammatory response during the acute phase of myocardial infarction after simvastatin withdrawal. Atherosclerosis. 2009 Nov;207(1):191-4. doi: 10.1016/j.atherosclerosis.2009.04.008. Epub 2009 Apr 17. PMID 19464010
- [Result] Quinaglia e Silva JC, Munhoz DB, Morato TN, Gurgel A, Macedo AC, Sever P, Sposito AC; Brasilia Heart Study Group. Effect of beta blockers (metoprolol or propranolol) on effect of simvastatin in lowering C-reactive protein in acute myocardial infarction. Am J Cardiol. 2009 Feb 15;103(4):461-3. doi: 10.1016/j.amjcard.2008.10.007. Epub 2008 Dec 25. PMID 19195502
- [Result] Carvalho LS, Virginio VW, Panzoldo NB, Figueiredo VN, Santos SN, Modolo RG, Andrade JM, Quinaglia E Silva JC, Nadruz-Junior W, de Faria EC, Sposito AC; Brasilia Heart Study Group. Elevated CETP activity during acute phase of myocardial infarction is independently associated with endothelial dysfunction and adverse clinical outcome. Atherosclerosis. 2014 Dec;237(2):777-83. doi: 10.1016/j.atherosclerosis.2014.10.104. Epub 2014 Nov 4. PMID 25463120
- [Result] Carvalho LS, Panzoldo N, Santos SN, Modolo R, Almeida B, Quinaglia E Silva JC, Nadruz W Jr, de Faria EC, Sposito AC; Brasilia Heart Study Group. HDL levels and oxidizability during myocardial infarction are associated with reduced endothelial-mediated vasodilation and nitric oxide bioavailability. Atherosclerosis. 2014 Dec;237(2):840-6. doi: 10.1016/j.atherosclerosis.2014.10.103. Epub 2014 Nov 4. PMID 25463131
- [Result] Machado-Silva W, Alfinito-Kreis R, Carvalho LS, Quinaglia-E-Silva JC, Almeida OL, Brito CJ, Ferreira AP, Cordova C, Sposito AC, Nobrega OT; Brasilia Heart Study Group. Endothelial nitric oxide synthase genotypes modulate peripheral vasodilatory properties after myocardial infarction. Gene. 2015 Sep 1;568(2):165-9. doi: 10.1016/j.gene.2015.05.042. Epub 2015 May 20. PMID 26002446
- [Result] Modolo R, Figueiredo VN, Moura FA, Almeida B, Quinaglia e Silva JC, Nadruz W Jr, Lemos PA, Coelho OR, Blaha MJ, Sposito AC; Brasilia Heart Study Group. Coronary artery calcification score is an independent predictor of the no-reflow phenomenon after reperfusion therapy in acute myocardial infarction. Coron Artery Dis. 2015 Nov;26(7):562-6. doi: 10.1097/MCA.0000000000000269. PMID 26010531
- [Derived] Barreto J, Matos LCV, Quinaglia JC, Sposito AC, Carvalho LS. The impact of low income on long-term mortality of myocardial infarction patients: results from the Brazilian Heart Study. Curr Med Res Opin. 2021 Oct;37(10):1689-1695. doi: 10.1080/03007995.2021.1965561. Epub 2021 Aug 17. PMID 34374619
- [Derived] Campos-Staffico AM, Costa APR, Carvalho LSF, Moura FA, Santos SN, Coelho-Filho OR, Nadruz W Jr, Quinaglia E Silva JC, Sposito AC; Brasilia Heart Study. Omega-3 intake is associated with attenuated inflammatory response and cardiac remodeling after myocardial infarction. Nutr J. 2019 May 6;18(1):29. doi: 10.1186/s12937-019-0455-1. PMID 31060562
- See also: Facebook page about the study. — https://www.facebook.com/Brazilian.Heart.Study